CLINICAL TRIAL: NCT06253715
Title: Shortened Regimen for Drug-susceptible TB in Children
Acronym: SMILE-TB
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00388853
Record Dates: First submitted 2024-01-26; First posted 2024-02-12 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary; Tuberculosis, Lymph Node; Mycobacterium Tuberculosis
Keywords: tuberculosis; pediatric; stratified medicine; shortened regimen; rifapentine; moxifloxacin; dolutegravir; drug-susceptible; lymph node; pulmonary; infections; TB; mycobacterium infections; respiratory tract infections; lung diseases; antitubercular agents; respiratory tract diseases; child; paediatric
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary; Tuberculosis, Lymph Node; Infections; Mycobacterium Infections; Respiratory Tract Infections; Lung Diseases; Respiratory Tract Diseases | interventions — Isoniazid; Protons; Rifampin; Pyrazinamide; Ethambutol; rifapentine; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: International, multicenter, randomized, controlled, open-label, non-inferiority
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regimen 1: Isoniazid (H), Rifampin (R), Pyrazinamide (Z), Ethambutol (E) (Active Comparator): 8 weeks of daily HRZ(E) followed by either 16 or 24 weeks of daily HR, per local standard of care
  Interventions: Drug: Isoniazid; Drug: Rifampin; Drug: Pyrazinamide; Drug: Ethambutol
- Regimen 2: Isoniazid (H), Rifapentine (P), Pyrazinamide (Z), Moxifloxacin (M) (Experimental): 8 weeks of daily HPZM
  Interventions: Drug: Isoniazid; Drug: Pyrazinamide; Drug: Rifapentine; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Isoniazid — Once daily weight-based dose
  Other Names: H
Drug: Rifampin — Once daily weight-based dose
  Other Names: R
  Arms: Regimen 1: Isoniazid (H), Rifampin (R), Pyrazinamide (Z), Ethambutol (E)
Drug: Pyrazinamide — Once daily weight-based dose
  Other Names: Z
Drug: Ethambutol — Once daily weight-based dose
  Other Names: E
  Arms: Regimen 1: Isoniazid (H), Rifampin (R), Pyrazinamide (Z), Ethambutol (E)
Drug: Rifapentine — Once daily weight-based dose
  Other Names: P; Priftin
  Arms: Regimen 2: Isoniazid (H), Rifapentine (P), Pyrazinamide (Z), Moxifloxacin (M)
Drug: Moxifloxacin — Once daily weight-based dose
  Other Names: M; Avelox
  Arms: Regimen 2: Isoniazid (H), Rifapentine (P), Pyrazinamide (Z), Moxifloxacin (M)

SUMMARY:
While drug-susceptible tuberculosis (TB) disease in children currently requires four to six months of treatment, most children may be able to be cured with a shorter treatment of more powerful drugs. Shorter treatment may be easier for children to tolerate and finish as well as ease caregiver strain from managing treatment side effects and supporting children over many months. The primary objective of this study is to evaluate if a 2-month regimen (including isoniazid (H), rifapentine (P), pyrazinamide (Z) and moxifloxacin (M)) is as safe and effective as a 4- to 6-month regimen (isoniazid, rifampicin (R), pyrazinamide, ethambutol (E)) in curing drug-susceptible TB disease in children under 10 years old. The study is also evaluating the safety of the HPZM in children with and without HIV.

DETAILED DESCRIPTION:
In previously untreated individuals with presumed drug-susceptible pulmonary and or peripheral lymph node TB treated with eight weeks of rifapentine, isoniazid, pyrazinamide and moxifloxacin (2HPZM), all given daily throughout, the proportion of participants who experience absence of cure (unsuccessful outcome) will not be inferior to that observed in participants who are treated with the standard regimen (eight weeks of rifampin, isoniazid, pyrazinamide, with or without ethambutol followed by 8 to 16 weeks of rifampin plus isoniazid depending on disease severity) all given daily throughout.

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian is willing and able to provide written informed consent for potential participant's study participation; in addition, when applicable per Ethics Committee/Institutional Review Board (EC/IRB) policies and procedures, potential participant is willing and able to provide assent for study participation.
* At Entry, age of less than 10 years.
* At Entry, weight 3 kilograms (kg) or greater.
* At Entry, diagnosed with TB disease, defined as:

  * Pulmonary (including pleural effusion) and/or lymph node (extra-thoracic and/or intra-thoracic) TB with or without bacteriologic confirmation;
  * Clinician has decided to treat with standard first-line drug-susceptible TB regimen.
* Known HIV status or HIV testing in progress based on meeting testing requirements.
* Has normal, Grade 1 or 2 test results for all of the following done at or within 14 days of Entry (including the most recent):

  * Alanine aminotransferase (ALT) less than or equal to 5 times the upper limit of normal;
  * Total bilirubin less than or equal to 2.5 times the upper limit of normal;
  * Potassium level of 3.0 milliequivalent/L or greater;
  * Hemoglobin level of 7.0 g/dL or greater;
  * Platelet count of 100,000/mm3 or greater;
  * Estimated glomerular filtration rate (eGFR; bedside Schwartz formula) 60 mL/min/1.73m2 or higher.
* For children living with HIV:

  * On antiretroviral therapy (ART) at Entry: Must be on, or able to be switched to a dolutegravir-based regimen at or prior to Entry;
  * Not on ART at Entry: Planned initiation of dolutegravir before or at study Week 4.
* For participants who have reached menarche or who are engaging in sexual activity (self-reported): negative serum or urine pregnancy test within 7 days of Entry.
* For participants who are engaging in sexual activity that could lead to pregnancy (self-reported): agrees to practice at least one non-hormonal method of contraception or abstain from heterosexual intercourse during study drug treatment and for 30 days after stopping study medications. Non-hormonal methods include:

  * Male or female condoms
  * Diaphragm or cervical cap (with spermicide, if available)
  * Non-hormonal intrauterine device (IUD) or intrauterine system (IUS)
* At Entry, intends to remain in the catchment area of the study site for the duration of study follow-up or willingness to be followed up beyond the catchment area if/when applicable, as determined by the site investigator based on participant/parent/guardian report.

Exclusion Criteria:

* Presumed or documented extra-pulmonary TB involving the central nervous system and/or bones and/or joints, and/or miliary TB, and/or pericardial TB and/or TB of the gastrointestinal (GI) tract and/or renal TB.
* Premature infant (born less than 37-weeks gestation) who is less than 3 months of age at Entry.
* Any known contraindication to taking any study drug:

  * Known allergy or intolerance to any of the study drugs or drugs in the same class as the study drugs;
  * Any prohibited medications within three days prior to Entry or planned use within the following 6 months;
  * Unable to take oral medications;
  * Known history of prolonged QT syndrome not caused by electrolyte derangements.
* Received more than 10 days of treatment directed against TB disease within 6 months preceding initiation of study drugs.
* M. tuberculosis isolate known or suspected to be resistant to isoniazid, rifampin, pyrazinamide, ethambutol, and/or fluoroquinolones.
* Known exposure to an infectious adult with drug-resistant TB, including resistance to isoniazid, rifampin, pyrazinamide, ethambutol, and/or fluoroquinolones.
* Has any other documented or suspected clinically significant medical condition or any other condition that, in the opinion of the site investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
* Previously enrolled in this study.

Late Exclusions:

* M. tuberculosis cultured or detected through World Health Organization (WHO) approved molecular assays (e.g., Cepheid Xpert MTB/RIF, Xpert XDR, sequencing or Hain MTB-DR plus assays) from sputum, swallowed sputum, nasopharyngeal aspirates, stool, or lymph node aspirate obtained around the time of study entry is determined to be resistant to isoniazid and/or rifampin and/or pyrazinamide and/or ethambutol and/or fluoroquinolones.
* Any child with a clinical TB diagnosis who is found to have a definitive alternative diagnosis for their presenting signs and symptoms whose TB treatment is discontinued prior to completion.

Ages: 0 Days to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 860 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
TB disease-free survival at 48-weeks | Measured from study entry through week 48
  Non-inferiority will be assessed by comparing the upper bound of a 95%, 2-sided confidence interval for the difference between the proportion of participants who are classified as having an unsuccessful outcome on the control regimen (HRZ(E)) and the intervention regimen (HPZM) to the predefined non-inferiority margin of 6% at 48 weeks.
Proportion of participants with grade 3 or higher adverse events over 28 weeks | Measured from study entry through Week 28
  The proportion of participants with a Grade 3 or higher adverse event and the corresponding 95% confidence intervals will be generated. An exact test for equality of proportions will be used to compare safety outcomes between the arms.

SECONDARY OUTCOMES:
TB disease-free survival at 48-weeks | Measured from study entry through Week 48
  Non-inferiority will be assessed by comparing the upper bound of a 95%, 2-sided confidence interval for the difference between the proportion of participants who are classified as having an unsuccessful outcome on the control regimen (HRZ(E)) and the intervention regimen (HPZM) to the predefined non-inferiority margin of 6% at 48 weeks.
TB disease-free survival at 72-weeks | Measured from study entry through Week 72
  Non-inferiority will be assessed by comparing the upper bound of a 95%, 2-sided confidence interval for the difference between the proportion of participants who are classified as having an unsuccessful outcome on the control regimen (HRZ(E)) and the intervention regimen (HPZM) to the predefined non-inferiority margin of 6% at 72 weeks.
Adherence to treatment regimens | Measured from study entry through Week 48
  The per-protocol analysis will account for variations in adherence to the treatment regimens. Inverse probability of treatment weighting (IPTW) using propensity scores will be applied and the net difference in treatment failure rates between the two treatment regimens and the 95% confidence interval around this will be calculated to determine non-inferiority.
Tolerability as assessed by proportion of participants who discontinue treatment | Week 8 (intervention/HPZM) or Week 16 or Week 24 (control/HRZ(E))
  Tolerability will be assessed as discontinuation of the assigned treatment for a reason other than microbiological ineligibility (AEs assessed as related to the study regimen that led to permanent discontinuation of the regimen, participant refusal, parent/guardian prematurely discontinues, etc.) among the modified intention-to-treat population. Proportion of participants who discontinue the assigned study regimen and the corresponding 95% confidence intervals will be generated. The control regimen (HRZ(E)) will be compared against the intervention regimen (HPZM) using an exact test for equality of proportions.
Rifapentine Area under the curve (AUC0-24) | Measured from study entry through Week 8
  Area under the curve from start of dose to 24 hours post-dose. Measured at Week 4 or Week 8. Blood samples drawn at 0, 1 minute, 2 minutes, 4 hours and 6 hours post dose.
Rifapentine minimal concentration (Cmin) | Measured from study entry through Week 8
  Minimal concentration from start of dose to 24 hours post-dose. Measured at Week 4 or Week 8. Blood samples drawn at 0, 1 minute, 2 minutes, 4 hours and 6 hours post dose.
Rifapentine peak concentration (Cmax) | Measured from study entry through Week 8
  Peak concentration from start of dose to 24 hours post-dose. Measured at Week 4 or Week 8. Blood samples drawn at 0, 1 minute, 2 minutes, 4 hours and 6 hours post dose.
Moxifloxacin AUC0-24 | Measured from study entry through Week 8
  Area under the curve from start of dose to 24 hours post-dose. Measured at Week 4 or Week 8. Blood samples drawn at 0, 1 minute, 2 minutes, 4 hours and 6 hours post dose.
Moxifloxacin Cmin | Measured from study entry through Week 8
  Minimal concentration from start of dose to 24 hours post-dose. Measured at Week 4 or Week 8. Blood samples drawn at 0, 1 minute, 2 minutes, 4 hours and 6 hours post dose.
Moxifloxacin Cmax | Measured from study entry through Week 8
  Peak concentration from start of dose to 24 hours post-dose. Measured at Week 4 or Week 8. Blood samples drawn at 0, 1 minute, 2 minutes, 4 hours and 6 hours post dose.
Parent/guardian and/or participant reported palatability and acceptability of study regimen | Baseline, Week 4, Week 8 (Regimens 1 and 2) and at Weeks 16 and 24 (Regimen 1 only)
  Based on questionnaire developed by study team, data will be aggregated to measure acceptability at Entry, Week 4, and Week 8 (all participants), and Weeks 16 and 24 (for those who continue on HRZ(E) only). Scoring based on a likert or likert-like scale for each question. Each question is scored 1 to 5 with higher scores reflecting increased acceptability.
Adherence as assessed by proportion of participants who have taken at least 90% of their doses | Baseline through Week 8 for HPZM, Week 16 for HRZ(E) with non-severe disease, or Week 24 for HRZ(E) with severe disease
  Adherence measures will be documented by a treatment supporter on a TB treatment card (as per local practice), by pill count and by an adherence questionnaire and descriptively summarized for all participants. Participants are considered adherent who have taken at least 90% of their doses within the 8 week, 16 week or 24-week time frame of their regimen.
Risk Stratification Algorithm | Measured from study entry through Week 48
  If the study outcome is not non-inferior, pragmatic, programmatically available data will be considered for inclusion in a risk stratification algorithm that would aim to identify children at high risk of unsuccessful TB treatment outcome who may benefit from a longer duration of therapy. The efficacy endpoint will be analyzed using mixed-effects logistic regression models to identify predictors. The models will be adjusted for World Bank country income categories and by site using random intercepts. Univariable and multivariable analysis will be performed. The association between baseline clinical predictors and unsuccessful treatment outcomes will be analyzed, Treatment characteristics will then be added to the models to determine if treatment helped in the description of the primary efficacy endpoint.
Cost effectiveness as assessed by the incremental cost-effective ratio (ICER) | Measured from study entry through Week 24
  ICER: Total costs of HPZM minus the total costs 16 or 24 week HRZE, divided by the total number of disability-adjusted life-year (DALY) averted for HPZM minus the total DALYs averted for 16- or 24-week HRZE.

OTHER OUTCOMES:
Dolutegravir AUC0-24 | Measured from study entry through Week 28
  Area under the curve from start of dose to 24 hours post-dose. Measured at Week 4 or 8 and at between Weeks 12-28. Blood samples drawn at 0, 1 hour, 4 hours and 6 hours post dose.
Dolutegravir Cmin | Measured from study entry through Week 28
  Minimal concentration from start of dose to 24 hours post-dose. Measured at Week 4 or 8 and at between Weeks 12-28. Blood samples drawn at 0, 1 hour, 4 hours and 6 hours post dose.
Dolutegravir Cmax | Measured from study entry through Week 28
  Peak concentration from start of dose to 24 hours post-dose. Measured at Week 4 or 8 and at between Weeks 12-28. Blood samples drawn at 0, 1 hour, 4 hours and 6 hours post dose.
Proportion of children living with HIV | Week 24 and Week 48
  Among participants living with HIV, the proportions of participants in each study arm who achieve or maintain virologic control (< 200 copies/mL) at Weeks 24 and 48 will be presented in aggregate, as well as broken down by weight bands (if the sample sizes are sufficient) bounded by 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Salazar-Austin, MD, ScM, Principal Investigator — Johns Hopkins University
Locations (9):
- India (2):
  - Indian Council of Medical Research - National Institute for Research in Tuberculosis, Chennai
  - Dr. D.Y. Patil Medical College, Hospital and Research Center, Pune
- Faculty of Medicine, Universitas Padjadjaran, Bandung, Indonesia
- Instituto Nacional de Saúde (INS), Maputo, Mozambique
- Africa Health Research Institute (AHRI), Durban, South Africa
- MU-JHU Care Ltd, Kampala, Uganda
- Zambia (2):
  - University of Zambia, School of Medicine, Lusaka
  - Arthur Davison Children's Hospital, Ndola
- Harare Health and Research Consortium (HHRC), Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Make individual participant data, after de-identification, publicly available in accordance with USAID's policy on data sharing.
Time Frame: After study completion, de-identified data that can be legally released to the public may be released.
Access Criteria: With whom: Researchers who provide a methodologically sound proposal for the use of the data per USAID's policy on data sharing and in accordance with in-country data sharing agreements.
  For what types of analysis: To achieve aims specified in the researcher's approved proposal.
  By what mechanisms will data be available: To be determined.

REFERENCES:
- [Background] Avelox package insert. U.S. Food and Drug Administration. (2016). Label: Avelox (moxifloxacin hydrochloride) tablets. URL: https://www.accessdata.fda.gov/drugsatfda_docs/label/2016/021085s063lbl.pdf
- [Background] Baciewicz AM, Self TH. Isoniazid interactions. South Med J. 1985 Jun;78(6):714-8. doi: 10.1097/00007611-198506000-00025. PMID 3890202
- [Background] Ball P. Moxifloxacin (Avelox): an 8-methoxyquinolone antibacterial with enhanced potency. Int J Clin Pract. 2000 Jun;54(5):329-32. PMID 10954961
- [Background] Berg A, Clary J, Hanna D, Nuermberger E, Lenaerts A, Ammerman N, Ramey M, Hartley D, Hermann D. Model-Based Meta-Analysis of Relapsing Mouse Model Studies from the Critical Path to Tuberculosis Drug Regimens Initiative Database. Antimicrob Agents Chemother. 2022 Mar 15;66(3):e0179321. doi: 10.1128/AAC.01793-21. Epub 2022 Jan 31. PMID 35099274
- [Background] Blumberg HM, Burman WJ, Chaisson RE, Daley CL, Etkind SC, Friedman LN, Fujiwara P, Grzemska M, Hopewell PC, Iseman MD, Jasmer RM, Koppaka V, Menzies RI, O'Brien RJ, Reves RR, Reichman LB, Simone PM, Starke JR, Vernon AA; American Thoracic Society, Centers for Disease Control and Prevention and the Infectious Diseases Society. American Thoracic Society/Centers for Disease Control and Prevention/Infectious Diseases Society of America: treatment of tuberculosis. Am J Respir Crit Care Med. 2003 Feb 15;167(4):603-62. doi: 10.1164/rccm.167.4.603. No abstract available. PMID 12588714
- [Background] Burman WJ, Goldberg S, Johnson JL, Muzanye G, Engle M, Mosher AW, Choudhri S, Daley CL, Munsiff SS, Zhao Z, Vernon A, Chaisson RE. Moxifloxacin versus ethambutol in the first 2 months of treatment for pulmonary tuberculosis. Am J Respir Crit Care Med. 2006 Aug 1;174(3):331-8. doi: 10.1164/rccm.200603-360OC. Epub 2006 May 4. PMID 16675781
- [Background] Centers for Disease Control and Prevention. (2023, March 22). Tuberculosis (TB) Treatment, Treatment for TB Disease. https://www.cdc.gov/tb/topic/treatment/tbdisease.htm
- [Background] Combs DL, O'Brien RJ, Geiter LJ. USPHS Tuberculosis Short-Course Chemotherapy Trial 21: effectiveness, toxicity, and acceptability. The report of final results. Ann Intern Med. 1990 Mar 15;112(6):397-406. doi: 10.7326/0003-4819-76-3-112-6-397. PMID 2155569
- [Background] Conde MB, Efron A, Loredo C, De Souza GR, Graca NP, Cezar MC, Ram M, Chaudhary MA, Bishai WR, Kritski AL, Chaisson RE. Moxifloxacin versus ethambutol in the initial treatment of tuberculosis: a double-blind, randomised, controlled phase II trial. Lancet. 2009 Apr 4;373(9670):1183-9. doi: 10.1016/S0140-6736(09)60333-0. PMID 19345831
- [Background] Donald PR, Maritz JS, Diacon AH. The pharmacokinetics and pharmacodynamics of rifampicin in adults and children in relation to the dosage recommended for children. Tuberculosis (Edinb). 2011 May;91(3):196-207. doi: 10.1016/j.tube.2011.02.004. Epub 2011 Mar 22. PMID 21429802
- [Background] Dooley KE, Park JG, Swindells S, Allen R, Haas DW, Cramer Y, Aweeka F, Wiggins I, Gupta A, Lizak P, Qasba S, van Heeswijk R, Flexner C; ACTG 5267 Study Team. Safety, tolerability, and pharmacokinetic interactions of the antituberculous agent TMC207 (bedaquiline) with efavirenz in healthy volunteers: AIDS Clinical Trials Group Study A5267. J Acquir Immune Defic Syndr. 2012 Apr 15;59(5):455-62. doi: 10.1097/QAI.0b013e3182410503. PMID 22126739
- [Background] Dooley KE, Bliven-Sizemore EE, Weiner M, Lu Y, Nuermberger EL, Hubbard WC, Fuchs EJ, Melia MT, Burman WJ, Dorman SE. Safety and pharmacokinetics of escalating daily doses of the antituberculosis drug rifapentine in healthy volunteers. Clin Pharmacol Ther. 2012 May;91(5):881-8. doi: 10.1038/clpt.2011.323. PMID 22472995
- [Background] Dooley KE, Kaplan R, Mwelase N, Grinsztejn B, Ticona E, Lacerda M, Sued O, Belonosova E, Ait-Khaled M, Angelis K, Brown D, Singh R, Talarico CL, Tenorio AR, Keegan MR, Aboud M; International Study of Patients with HIV on Rifampicin ING study group. Dolutegravir-based Antiretroviral Therapy for Patients Coinfected With Tuberculosis and Human Immunodeficiency Virus: A Multicenter, Noncomparative, Open-label, Randomized Trial. Clin Infect Dis. 2020 Feb 3;70(4):549-556. doi: 10.1093/cid/ciz256. PMID 30918967
- [Background] Dorman SE, Goldberg S, Stout JE, Muzanyi G, Johnson JL, Weiner M, Bozeman L, Heilig CM, Feng PJ, Moro R, Narita M, Nahid P, Ray S, Bates E, Haile B, Nuermberger EL, Vernon A, Schluger NW; Tuberculosis Trials Consortium. Substitution of rifapentine for rifampin during intensive phase treatment of pulmonary tuberculosis: study 29 of the tuberculosis trials consortium. J Infect Dis. 2012 Oct 1;206(7):1030-40. doi: 10.1093/infdis/jis461. Epub 2012 Jul 30. PMID 22850121
- [Background] Dorman SE, Savic RM, Goldberg S, Stout JE, Schluger N, Muzanyi G, Johnson JL, Nahid P, Hecker EJ, Heilig CM, Bozeman L, Feng PJ, Moro RN, MacKenzie W, Dooley KE, Nuermberger EL, Vernon A, Weiner M; Tuberculosis Trials Consortium. Daily rifapentine for treatment of pulmonary tuberculosis. A randomized, dose-ranging trial. Am J Respir Crit Care Med. 2015 Feb 1;191(3):333-43. doi: 10.1164/rccm.201410-1843OC. PMID 25489785
- [Background] Dorman SE, Nahid P, Kurbatova EV, Goldberg SV, Bozeman L, Burman WJ, Chang KC, Chen M, Cotton M, Dooley KE, Engle M, Feng PJ, Fletcher CV, Ha P, Heilig CM, Johnson JL, Lessem E, Metchock B, Miro JM, Nhung NV, Pettit AC, Phillips PPJ, Podany AT, Purfield AE, Robergeau K, Samaneka W, Scott NA, Sizemore E, Vernon A, Weiner M, Swindells S, Chaisson RE; AIDS Clinical Trials Group and the Tuberculosis Trials Consortium. High-dose rifapentine with or without moxifloxacin for shortening treatment of pulmonary tuberculosis: Study protocol for TBTC study 31/ACTG A5349 phase 3 clinical trial. Contemp Clin Trials. 2020 Mar;90:105938. doi: 10.1016/j.cct.2020.105938. Epub 2020 Jan 22. PMID 31981713
- [Background] Dorman SE, Nahid P, Kurbatova EV, Phillips PPJ, Bryant K, Dooley KE, Engle M, Goldberg SV, Phan HTT, Hakim J, Johnson JL, Lourens M, Martinson NA, Muzanyi G, Narunsky K, Nerette S, Nguyen NV, Pham TH, Pierre S, Purfield AE, Samaneka W, Savic RM, Sanne I, Scott NA, Shenje J, Sizemore E, Vernon A, Waja Z, Weiner M, Swindells S, Chaisson RE; AIDS Clinical Trials Group; Tuberculosis Trials Consortium. Four-Month Rifapentine Regimens with or without Moxifloxacin for Tuberculosis. N Engl J Med. 2021 May 6;384(18):1705-1718. doi: 10.1056/NEJMoa2033400. PMID 33951360
- [Background] Dossing M, Wilcke JT, Askgaard DS, Nybo B. Liver injury during antituberculosis treatment: an 11-year study. Tuber Lung Dis. 1996 Aug;77(4):335-40. doi: 10.1016/s0962-8479(96)90098-2. PMID 8796249
- [Background] Ellard GA. Absorption, metabolism and excretion of pyrazinamide in man. Tubercle. 1969 Jun;50(2):144-58. doi: 10.1016/0041-3879(69)90020-8. No abstract available. PMID 5788407
- [Background] Ellard GA. The potential clinical significance of the isoniazid acetylator phenotype in the treatment of pulmonary tuberculosis. Tubercle. 1984 Sep;65(3):211-27. doi: 10.1016/0041-3879(84)90079-5. No abstract available. PMID 6385429
- [Background] Ellard GA, Humphries MJ, Gabriel M, Teoh R. Penetration of pyrazinamide into the cerebrospinal fluid in tuberculous meningitis. Br Med J (Clin Res Ed). 1987 Jan 31;294(6567):284-5. doi: 10.1136/bmj.294.6567.284. No abstract available. PMID 3101843
- [Background] Food and Drug Administration (FDA). Guidance on General Clinical Pharmacology Considerations for Pediatric Studies for Drugs and Biological Products: Guidance for Industry (draft guidance) December 2014. [Available from: https://www.fda.gov/media/90358/download.]
- [Background] Gillespie SH, Crook AM, McHugh TD, Mendel CM, Meredith SK, Murray SR, Pappas F, Phillips PP, Nunn AJ; REMoxTB Consortium. Four-month moxifloxacin-based regimens for drug-sensitive tuberculosis. N Engl J Med. 2014 Oct 23;371(17):1577-87. doi: 10.1056/NEJMoa1407426. Epub 2014 Sep 7. PMID 25196020
- [Background] Griesel R, Hill A, Meintjes G, Maartens G. Standard versus double dose dolutegravir in patients with HIV-associated tuberculosis: a phase 2 non-comparative randomised controlled (RADIANT-TB) trial. Wellcome Open Res. 2021 Jan 11;6:1. doi: 10.12688/wellcomeopenres.16473.1. eCollection 2021. PMID 33954265
- [Background] Griesel R, Zhao Y, Simmons B, Omar Z, Wiesner L, Keene CM, Hill AM, Meintjes G, Maartens G. Standard-dose versus double-dose dolutegravir in HIV-associated tuberculosis in South Africa (RADIANT-TB): a phase 2, non-comparative, randomised controlled trial. Lancet HIV. 2023 Jul;10(7):e433-e441. doi: 10.1016/S2352-3018(23)00081-4. Epub 2023 May 22. PMID 37230101
- [Background] Hibma JE, Radtke KK, Dorman SE, Jindani A, Dooley KE, Weiner M, McIlleron HM, Savic RM. Rifapentine Population Pharmacokinetics and Dosing Recommendations for Latent Tuberculosis Infection. Am J Respir Crit Care Med. 2020 Sep 15;202(6):866-877. doi: 10.1164/rccm.201912-2489OC. PMID 32412342
- [Background] Hsu AJ, Tamma PD. The Johns Hopkins Hospital Antibiotics Guidelines 2023-2024. Treatment recommendations for hospitalized children. 2022 Johns Hopkins Medicine. Website: https://intranet.insidehopkinsmedicine.org/asp/pediatric.html. Last visited on: October 9th, 2023.
- [Background] Imperial MZ, Luetkenmeyer A, Dawson R, et al; the ACTG A5372 Protocol Team. DTG PK In People With HIV Receiving Daily 1HP For Latent TB Treatment (ACTG A5372). CROI, Conference on Retroviruses and Opportunistic Infections, 2022, Feb 15. Abstract 78.
- [Background] Jindani A, Harrison TS, Nunn AJ, Phillips PP, Churchyard GJ, Charalambous S, Hatherill M, Geldenhuys H, McIlleron HM, Zvada SP, Mungofa S, Shah NA, Zizhou S, Magweta L, Shepherd J, Nyirenda S, van Dijk JH, Clouting HE, Coleman D, Bateson AL, McHugh TD, Butcher PD, Mitchison DA; RIFAQUIN Trial Team. High-dose rifapentine with moxifloxacin for pulmonary tuberculosis. N Engl J Med. 2014 Oct 23;371(17):1599-608. doi: 10.1056/NEJMoa1314210. PMID 25337749
- [Background] Kay L, Kampmann JP, Svendsen TL, Vergman B, Hansen JE, Skovsted L, Kristensen M. Influence of rifampicin and isoniazid on the kinetics of phenytoin. Br J Clin Pharmacol. 1985 Oct;20(4):323-6. doi: 10.1111/j.1365-2125.1985.tb05071.x. PMID 4074601
- [Background] Kjellsson MC, Via LE, Goh A, Weiner D, Low KM, Kern S, Pillai G, Barry CE 3rd, Dartois V. Pharmacokinetic evaluation of the penetration of antituberculosis agents in rabbit pulmonary lesions. Antimicrob Agents Chemother. 2012 Jan;56(1):446-57. doi: 10.1128/AAC.05208-11. Epub 2011 Oct 10. PMID 21986820
- [Background] Kohno S, Koga H, Kaku M, Maesaki S, Hara K. Prospective comparative study of ofloxacin or ethambutol for the treatment of pulmonary tuberculosis. Chest. 1992 Dec;102(6):1815-8. doi: 10.1378/chest.102.6.1815. PMID 1446494
- [Background] Lacroix C, Tranvouez JL, Phan Hoang T, Duwoos H, Lafont O. Pharmacokinetics of pyrazinamide and its metabolites in patients with hepatic cirrhotic insufficiency. Arzneimittelforschung. 1990 Jan;40(1):76-9. PMID 2340003
- [Background] Mathad JS, Queiroz ATL, Bhosale R, Alexander M, Naik S, Kulkarni V, Andrade BB, Gupta A. Transcriptional Analysis for Tuberculosis in Pregnant Women From the PRegnancy Associated Changes In Tuberculosis Immunology (PRACHITi) Study. Clin Infect Dis. 2022 Dec 19;75(12):2239-2242. doi: 10.1093/cid/ciac437. PMID 35686302
- [Background] Merle CS, Fielding K, Sow OB, Gninafon M, Lo MB, Mthiyane T, Odhiambo J, Amukoye E, Bah B, Kassa F, N'Diaye A, Rustomjee R, de Jong BC, Horton J, Perronne C, Sismanidis C, Lapujade O, Olliaro PL, Lienhardt C; OFLOTUB/Gatifloxacin for Tuberculosis Project. A four-month gatifloxacin-containing regimen for treating tuberculosis. N Engl J Med. 2014 Oct 23;371(17):1588-98. doi: 10.1056/NEJMoa1315817. PMID 25337748
- [Background] Moro RN, Scott NA, Vernon A, Tepper NK, Goldberg SV, Schwartzman K, Leung CC, Schluger NW, Belknap RW, Chaisson RE, Narita M, Machado ES, Lopez M, Sanchez J, Villarino ME, Sterling TR. Exposure to Latent Tuberculosis Treatment during Pregnancy. The PREVENT TB and the iAdhere Trials. Ann Am Thorac Soc. 2018 May;15(5):570-580. doi: 10.1513/AnnalsATS.201704-326OC. PMID 29393655
- [Background] Ormerod LP, Horsfield N. Frequency and type of reactions to antituberculosis drugs: observations in routine treatment. Tuber Lung Dis. 1996 Feb;77(1):37-42. doi: 10.1016/s0962-8479(96)90073-8. PMID 8733412
- [Background] Bemer-Melchior P, Bryskier A, Drugeon HB. Comparison of the in vitro activities of rifapentine and rifampicin against Mycobacterium tuberculosis complex. J Antimicrob Chemother. 2000 Oct;46(4):571-6. doi: 10.1093/jac/46.4.571. PMID 11020254
- [Background] Patel AM, McKeon J. Avoidance and management of adverse reactions to antituberculosis drugs. Drug Saf. 1995 Jan;12(1):1-25. doi: 10.2165/00002018-199512010-00001. PMID 7741981
- [Background] Patel K, Goldman JL. Safety Concerns Surrounding Quinolone Use in Children. J Clin Pharmacol. 2016 Sep;56(9):1060-75. doi: 10.1002/jcph.715. Epub 2016 Mar 28. PMID 26865283
- [Background] Peloquin CA, Namdar R, Dodge AA, Nix DE. Pharmacokinetics of isoniazid under fasting conditions, with food, and with antacids. Int J Tuberc Lung Dis. 1999 Aug;3(8):703-10. PMID 10460103
- [Background] Pierfitte C, Royer RJ. Tendon disorders with fluoroquinolones. Therapie. 1996 Jul-Aug;51(4):419-20. No abstract available. PMID 8953821
- [Background] Prideaux B, Dartois V, Staab D, Weiner DM, Goh A, Via LE, Barry CE 3rd, Stoeckli M. High-sensitivity MALDI-MRM-MS imaging of moxifloxacin distribution in tuberculosis-infected rabbit lungs and granulomatous lesions. Anal Chem. 2011 Mar 15;83(6):2112-8. doi: 10.1021/ac1029049. Epub 2011 Feb 18. PMID 21332183
- [Background] Priftin package insert. National Institute of Allergy and Infectious Diseases. (2021, July). Rifapentine (Priftin) Prescribing Information. National Institute of Allergy and Infectious Diseases.https://rsc.niaid.nih.gov/sites/default/files/Rifapentine%20%28Priftin%29%20PI_dated%20July%202021.pdf
- [Background] Radtke KK, Hesseling AC, Winckler JL, Draper HR, Solans BP, Thee S, Wiesner L, van der Laan LE, Fourie B, Nielsen J, Schaaf HS, Savic RM, Garcia-Prats AJ. Moxifloxacin Pharmacokinetics, Cardiac Safety, and Dosing for the Treatment of Rifampicin-Resistant Tuberculosis in Children. Clin Infect Dis. 2022 Apr 28;74(8):1372-1381. doi: 10.1093/cid/ciab641. PMID 34286843
- [Background] Reves R, Heilig CM, Tapy JM, Bozeman L, Kyle RP, Hamilton CD, Bock N, Narita M, Wing D, Hershfield E, Goldberg SV; Tuberculosis Trials Consortium. Intermittent tuberculosis treatment for patients with isoniazid intolerance or drug resistance. Int J Tuberc Lung Dis. 2014 May;18(5):571-80. doi: 10.5588/ijtld.13.0304. PMID 24903795
- [Background] Rosenthal IM, Zhang M, Williams KN, Peloquin CA, Tyagi S, Vernon AA, Bishai WR, Chaisson RE, Grosset JH, Nuermberger EL. Daily dosing of rifapentine cures tuberculosis in three months or less in the murine model. PLoS Med. 2007 Dec;4(12):e344. doi: 10.1371/journal.pmed.0040344. PMID 18092886
- [Background] Rosenthal IM, Zhang M, Almeida D, Grosset JH, Nuermberger EL. Isoniazid or moxifloxacin in rifapentine-based regimens for experimental tuberculosis? Am J Respir Crit Care Med. 2008 Nov 1;178(9):989-93. doi: 10.1164/rccm.200807-1029OC. Epub 2008 Aug 21. PMID 18723432
- [Background] Rosenthal IM, Tasneen R, Peloquin CA, Zhang M, Almeida D, Mdluli KE, Karakousis PC, Grosset JH, Nuermberger EL. Dose-ranging comparison of rifampin and rifapentine in two pathologically distinct murine models of tuberculosis. Antimicrob Agents Chemother. 2012 Aug;56(8):4331-40. doi: 10.1128/AAC.00912-12. Epub 2012 Jun 4. PMID 22664964
- [Background] Rustomjee R, Lienhardt C, Kanyok T, Davies GR, Levin J, Mthiyane T, Reddy C, Sturm AW, Sirgel FA, Allen J, Coleman DJ, Fourie B, Mitchison DA; Gatifloxacin for TB (OFLOTUB) study team. A Phase II study of the sterilising activities of ofloxacin, gatifloxacin and moxifloxacin in pulmonary tuberculosis. Int J Tuberc Lung Dis. 2008 Feb;12(2):128-38. PMID 18230244
- [Background] Sanofi. Rifadin [rifampin] package insert. Sanofi. 2023, February. URL:https://products.sanofi.us/rifadin/rifadin.pdf.
- [Background] Schaberg T, Rebhan K, Lode H. Risk factors for side-effects of isoniazid, rifampin and pyrazinamide in patients hospitalized for pulmonary tuberculosis. Eur Respir J. 1996 Oct;9(10):2026-30. doi: 10.1183/09031936.96.09102026. PMID 8902462
- [Background] Seddon JA, Garcia-Prats AJ, Purchase SE, Osman M, Demers AM, Hoddinott G, Crook AM, Owen-Powell E, Thomason MJ, Turkova A, Gibb DM, Fairlie L, Martinson N, Schaaf HS, Hesseling AC. Levofloxacin versus placebo for the prevention of tuberculosis disease in child contacts of multidrug-resistant tuberculosis: study protocol for a phase III cluster randomised controlled trial (TB-CHAMP). Trials. 2018 Dec 20;19(1):693. doi: 10.1186/s13063-018-3070-0. PMID 30572905
- [Background] Segev S, Yaniv I, Haverstock D, Reinhart H. Safety of long-term therapy with ciprofloxacin: data analysis of controlled clinical trials and review. Clin Infect Dis. 1999 Feb;28(2):299-308. doi: 10.1086/515132. PMID 10064248
- [Background] Snider DE Jr. Pyridoxine supplementation during isoniazid therapy. Tubercle. 1980 Dec;61(4):191-6. doi: 10.1016/0041-3879(80)90038-0. PMID 6269259
- [Background] Turkova A, Wills GH, Wobudeya E, Chabala C, Palmer M, Kinikar A, Hissar S, Choo L, Musoke P, Mulenga V, Mave V, Joseph B, LeBeau K, Thomason MJ, Mboizi RB, Kapasa M, van der Zalm MM, Raichur P, Bhavani PK, McIlleron H, Demers AM, Aarnoutse R, Love-Koh J, Seddon JA, Welch SB, Graham SM, Hesseling AC, Gibb DM, Crook AM; SHINE Trial Team. Shorter Treatment for Nonsevere Tuberculosis in African and Indian Children. N Engl J Med. 2022 Mar 10;386(10):911-922. doi: 10.1056/NEJMoa2104535. PMID 35263517
- [Background] Turkova A, Waalewijn H, Chan MK, Bollen PDJ, Bwakura-Dangarembizi MF, Kekitiinwa AR, Cotton MF, Lugemwa A, Variava E, Ahimbisibwe GM, Srirompotong U, Mumbiro V, Amuge P, Zuidewind P, Ali S, Kityo CM, Archary M, Ferrand RA, Violari A, Gibb DM, Burger DM, Ford D, Colbers A; ODYSSEY Trial Team. Dolutegravir twice-daily dosing in children with HIV-associated tuberculosis: a pharmacokinetic and safety study within the open-label, multicentre, randomised, non-inferiority ODYSSEY trial. Lancet HIV. 2022 Sep;9(9):e627-e637. doi: 10.1016/S2352-3018(22)00160-6. Epub 2022 Jul 19. PMID 35868341
- [Background] UNAIDS. (2022, March 24). Fact Sheet - Tuberculosis (TB) and HIV. https://www.unaids.org/sites/default/files/media_asset/20220324_TB_FactSheet_en.pdf
- [Background] Weiner M, Savic RM, Kenzie WR, Wing D, Peloquin CA, Engle M, Bliven E, Prihoda TJ, Gelfond JA, Scott NA, Abdel-Rahman SM, Kearns GL, Burman WJ, Sterling TR, Villarino ME; Tuberculosis Trials Consortium PREVENT TB Pharmacokinetic Group. Rifapentine Pharmacokinetics and Tolerability in Children and Adults Treated Once Weekly With Rifapentine and Isoniazid for Latent Tuberculosis Infection. J Pediatric Infect Dis Soc. 2014 Jun;3(2):132-45. doi: 10.1093/jpids/pit077. Epub 2014 Jan 16. PMID 26625366
- [Background] Williamson B, Dooley KE, Zhang Y, Back DJ, Owen A. Induction of influx and efflux transporters and cytochrome P450 3A4 in primary human hepatocytes by rifampin, rifabutin, and rifapentine. Antimicrob Agents Chemother. 2013 Dec;57(12):6366-9. doi: 10.1128/AAC.01124-13. Epub 2013 Sep 23. PMID 24060875
- [Background] Wirth S, Emil SGS, Engelis A, Digtyar V, Criollo M, DiCasoli C, Stass H, Willmann S, Nkulikiyinka R, Grossmann U; MOXIPEDIA Study Group. Moxifloxacin in Pediatric Patients With Complicated Intra-abdominal Infections: Results of the MOXIPEDIA Randomized Controlled Study. Pediatr Infect Dis J. 2018 Aug;37(8):e207-e213. doi: 10.1097/INF.0000000000001910. PMID 29356761
- [Background] World Health Organization, Global Tuberculosis Programme, Maternal, Newborn, Child & Adolescent Health & Ageing (2006). Ethambutol efficacy and toxicity: literature review and recommendations for daily and intermittent dosage in children. WHO/HTM/TB/2006.365, WHO/FCH/CAH/2006.3.
- [Background] World Health Organization (WHO), and UNITAID. Toolkit for research and development of paediatric antiretroviral drugs and formulations. Geneva: World Health Organization; 2018. License: CC BY-NC-SA 3.0 IGO. URL: https://iris.who.int/bitstream/handle/10665/273151/9789241514361-eng.pdf?sequence=1
- [Background] World Health Organization (2022a) WHO Global Tuberculosis Report 2022. Global Tuberculosis Programme, Tuberculosis Vaccine Accelerator Council. October, 2022. ISBN: 978-92-4-006172-9.
- [Background] WHO consolidated guidelines on tuberculosis: Module 4: Treatment - Drug-susceptible tuberculosis treatment [Internet]. Geneva: World Health Organization; 2022. Available from http://www.ncbi.nlm.nih.gov/books/NBK581329/ PMID 35727905
- [Background] WHO consolidated guidelines on tuberculosis: Module 5: Management of tuberculosis in children and adolescents [Internet]. Geneva: World Health Organization; 2022. Available from http://www.ncbi.nlm.nih.gov/books/NBK579387/ PMID 35404556
- [Background] World Health Organization (2022). Growth reference data for 5-19 years. [April 19, 2022]. Available from: https://www.who.int/tools/growth-reference-data-for-5to19-years.
- [Background] World Health Organization (2022). Child growth standards. [April 19, 2022]. Available from: https://www.who.int/tools/child-growth-standards.
- [Background] World Health Organization (2022f). Global Tuberculosis Report 2022; 3.3 TB treatment and treatment coverage. https://www.who.int/teams/global-tuberculosis-programme/tb-reports/global-tuberculosis-report-2022/tb-diagnosis-treatment/3-3-tb-treatment-and-treatment-coverage. Last visited: November 1, 2023.
- [Background] Yee D, Valiquette C, Pelletier M, Parisien I, Rocher I, Menzies D. Incidence of serious side effects from first-line antituberculosis drugs among patients treated for active tuberculosis. Am J Respir Crit Care Med. 2003 Jun 1;167(11):1472-7. doi: 10.1164/rccm.200206-626OC. Epub 2003 Jan 31. PMID 12569078
- [Background] Zent C, Smith P. Study of the effect of concomitant food on the bioavailability of rifampicin, isoniazid and pyrazinamide. Tuber Lung Dis. 1995 Apr;76(2):109-13. doi: 10.1016/0962-8479(95)90551-0. PMID 7780091
- [Background] Zhang T, Li SY, Williams KN, Andries K, Nuermberger EL. Short-course chemotherapy with TMC207 and rifapentine in a murine model of latent tuberculosis infection. Am J Respir Crit Care Med. 2011 Sep 15;184(6):732-7. doi: 10.1164/rccm.201103-0397OC. Epub 2011 Jun 9. PMID 21659613
- [Background] Zierski M, Bek E. Side-effects of drug regimens used in short-course chemotherapy for pulmonary tuberculosis. A controlled clinical study. Tubercle. 1980 Mar;61(1):41-9. doi: 10.1016/0041-3879(80)90060-4. PMID 6989067
- [Background] Zvada SP, Van Der Walt JS, Smith PJ, Fourie PB, Roscigno G, Mitchison D, Simonsson US, McIlleron HM. Effects of four different meal types on the population pharmacokinetics of single-dose rifapentine in healthy male volunteers. Antimicrob Agents Chemother. 2010 Aug;54(8):3390-4. doi: 10.1128/AAC.00345-10. Epub 2010 Jun 1. PMID 20516273